CLINICAL TRIAL: NCT04361448
Title: Comparison of the Performance of 3 Sampling Methods for the Detection of SARS-CoV-2 (COVID-19) With Real-time Reverse Transcriptase PCR
Brief Title: Performance of 3 Sampling Methods for the Detection of SARS-CoV-2 (COVID-19) With Real-time Reverse Transcriptase PCR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient sample number
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Reinoud Cartuyvels, MD, Jessa Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20.43
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Covid-19; SARS-CoV-2; Diagnosis; Polymerase Chain Reaction
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Intervention Model Description: Beside the regular sampling method of 1 nasopharyngeal swab, 2 extra swabs will be taken in each volunteer. Performance of the 3 methods for laboratory diagnosis by PCR of Covid-19 will be compared.
Masking Description: Each participant get study number. Samples will be identified by the study number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Care Workers with Covid-19 symptoms (Other): 3 samples (2 nasopharyngeasl swabs, 1 oropharyngeal swab) willl be taken from each volunteer
  Interventions: Other: samling of oropharynx and nasopharynx

INTERVENTIONS:
Other: samling of oropharynx and nasopharynx — Three different swabs will be taken of each participant: 1 oropharyngeal swab and 2 nasopharyngeal swabs

SUMMARY:
The performance of 3 different sampling methods (2 nasopharyngeal swabs, 1 oropharyngeal swab) for the detection of SARS-CoV-2 with real-time reverse transcriptase polymerase chain reaction will be compared.

DETAILED DESCRIPTION:
Thirty volunteers will be recruited from health care workers suspicious for Covid-19, who consult the ocupational physician for Covid-19 testing.

For each volunteer, 3 swabs will be taken:

* Flocked eSwab (Copan, Italy) of the oropharynx
* Flocked nasopharyngeal eSwab (Copan, Italy) of the nasopharynx
* Dry flocked nasopharyngeal Swab, placed in lysis buffer Each swab will be tested for the presence of SARS-CoV-2 with an in-house reverse-transcriptase real-time PCR (Egene).

Performance of each method will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* health care workers with symptoms suspicious for Covid-19

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
sensitivity | 1 month
  sensitivity of each sampling method for the detection of SARS-CoV-2 by RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Reinoud Cartuyvels, Principal Investigator — Jessa Hospital, Hasselt, Belgium
Locations (1):
- Jessa Hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No